CLINICAL TRIAL: NCT04263025
Title: Prospective, Controlled Study Evaluating Recovery of Potency and Continence Following Robot-Assisted Radical Prostatectomy With and Without Cryopreserved Umbilical Cord Allograft
Brief Title: AMNIOX CORD Study - Radical Prostatectomy With and Without Cryopreserved Umbilical Cord Allograft
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2019-0452
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Bilateral, nerve-sparing prostatectomy; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will be Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CLARIX CORD 1K (Experimental): They will receive adjunctive CLARIX® CORD 1K (Amniox Medical, Inc., Miami, FL) during Robot-Assisted Radical Prostatectomy (RARP).
  Interventions: Biological: Cryopreserved Umbilical Cord Allograft; Procedure: Robot-Assisted Radical Prostatectomy
- Controls (Active Comparator): They will undergo RARP without adjunctive CLARIX® CORD 1K.
  Interventions: Procedure: Robot-Assisted Radical Prostatectomy

INTERVENTIONS:
Biological: Cryopreserved Umbilical Cord Allograft — CLARIX® CORD 1K (Amniox Medical, Miami, FL) is an umbilical cord allograft processed using the patented CRYOTEK™ process by TissueTech Inc. to devitalize all living cells but retain the natural structural and biological characteristics relevant to this tissue [43]. CLARIX® CORD 1K (6x3 cm in size) will be cut into two longitudinal pieces (1.5 cm in width) and placed circumferentially around each NVB as a nerve wrap during RARP. CLARIX® CORD 1K has been in market since 2013 in the United States as a "361 human cell and tissue-based product (HCT/P)" and is aseptically processed in compliance with current Good Tissue Practices (cGTP) as outlined in 21 CFR Part 1271.
  Arms: CLARIX CORD 1K
Procedure: Robot-Assisted Radical Prostatectomy — Robot-Assisted Radical Prostatectomy (RARP) is the most common surgical technique used to treat clinically localized prostate cancer however robot-assisted radical prostatectomy

SUMMARY:
This study aims at evaluating if placement of CLARIX® CORD 1K during robotic prostatectomy decreases the time to achieve complete erectile and urinary function after the surgery. As part of the study, the patient will be asked to answer various questions after the surgery regarding sexual and urinary function.

DETAILED DESCRIPTION:
One hundred male patients who are scheduled for bilateral, nerve-sparing RARP that meet the eligibility criteria will be enrolled. These patients will be equally randomized (1:1) into two groups (n=50/group): one group will receive adjunctive CLARIX® CORD 1K (Amniox Medical, Inc., Miami, FL) during RARP, while the other group will undergo RARP without adjunctive CLARIX® CORD 1K. Subject stratification will be performed based on the surgeon that will be performing the RARP. All patients will be given the same routine preoperative, perioperative and postoperative evaluation and care aside from the CLARIX CORD 1K placement in the treatment group during RARP. RARP will be performed at Hackensack University Medical Center (30 Prospect Ave, Hackensack, NJ 07601) and follow up visits performed at Hackensack University Medical Group Urology (360 Essex Street, Suite 403, Hackensack, NJ 07601) or New Jersey Urology (255 W. Spring Valley Avenue Suite 101, Maywood, NJ 07607).

Two weeks prior to the RARP surgery, subjects are instructed to take low-dose oral phosphodiesterase type 5 inhibitors (i.e. 20 mg q.d. sildenafil citrate or 5 mg q.d. tadalafil) and perform standardized Kegel exercises (3x/day) which is our current standard care protocol. RARP surgery will be performed at Hackensack University Medical Center (Hackensack, NJ). The following are the key aspects of the RARP surgical technique which will be adhered to by all surgeons: 1) dissection of the bladder neck, seminal vesicles and vasa deferentia; 2) dissection of the neuroplexus from the posterior Denonvilliers' fascia and lateral prostatic fascia leaving the nerves intact; 3) division of the prostatic pedicles without cautery; 4) transection of the dorsal venous complex; and 5) urethrovesical anastomosis. More specifically, surgical technique includes exposing the prostate in the space of Retzius with the traditional anterior approach.

The prostatovesical tissue is dissected with monopolar electrocautery scissors with entry into the bladder proximal to the prostatovesical junction. The bladder neck is transected in the standard fashion followed by posterior dissection of the seminal vesicles and vasa deferentia.

Electrocautery is kept to a minimum when dissecting the seminal vesicles to avoid damage to the neuroplexus. (Note: each step hereafter must be performed by the PI or Sub-investigators, e.g. not a Resident Physician). A posterior surgical plane is then created between the rectum and prostate dorsally working from a medial to lateral direction and maintaining at least 1 layer of Denonvilliers' fascia on the rectal wall. The endopelvic fascia is then excised from lateral prostate and carried to capsule to create a plane of dissection immediately alongside the prostatic capsule and keeping the nerves attached laterally to the endopelvic fascia. Athermal division of each prostatic pedicle will be performed. Clips or suture may be placed on each pedicle at the discretion of the surgeon. The apex of the prostate is then dissected athermally sparing the neuroplexus. The dorsal vein complex is proximally transected with electrocautery while using the fourth arm to place traction on the prostate to define the space between the dorsal vein complex and the apex of the prostate. Apically, the prostate is divided from the urethra (paying special attention to the sphincter muscle and posterior lateral nerve bundle on each side) allowing the prostate to be removed. Once free, the prostate is placed in a collection bag and a drain is used for a certain period at the discretion of the surgeon.

Surgical site bleeding is managed using standard surgical techniques with sutures or cellulose polymer. If the patient is randomized to the treatment group, CLARIX CORD 1K is placed flat over the neuroplexis at the 5 and 7 clock position where the largest concentration of nerves exist. Sutures may be used to secure the CLARIX in place if necessary and cellulose polymer (Surgicel, Ethicon, Somerville, NJ) can be placed over the CLARIX CORD at the discretion of the physician.

At this point the bladder neck will be reconstructed as necessary to maintain a lumen of approximately 30 french. The vesicourethral anastomosis is performed using a V-lock barbed suture. The anastomosis will be tested by filling bladder to confirm the absence of leakage. If indicated, a bilateral pelvic lymph node dissection is performed (with clips at the discretion of the physician) using standard (borders along the external iliac artery and vein, obturator fossa, obturator nerve and pubic bone) or extended (borders additionally include internal iliac artery) technique at the discretion of the physician. Bleeding will be adequately managed. Postoperatively, all subjects are instructed to take low-dose oral phosphodiesterase type 5 inhibitors (i.e. 20 mg q.d. sildenafil citrate or 5 mg q.d. tadalafil) and perform standardized Kegel exercises (3x/day) following urethral catheter removal. When patients are sexually active, they may increase to full dosage of oral phosphodiesterase type 5 inhibitors up to twice a week. At 3 months after RARP, and if patients have severe or worse incontinence (defined as ICIQ score of >12) and desire additional treatment for urinary incontinence,[42] they will undergo pelvic floor therapy. Subjects will return for follow up visits at 6 weeks (±1 week), 3 months (±2 weeks), 6 months (±3 weeks) and 12 months (±4 weeks) when data will be collected.

Patient reported outcomes will be assessed including continence, potency, and satisfaction. Occurrence of adverse events, number of readmissions, and need for reintervention will also be recorded. Measurement of serum PSA levels will also be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged between 30 and 70 years old
2. Primary diagnosis of organ confined prostate cancer
3. Scheduled to undergo bilateral, nerve-sparing RARP
4. Patient has ICIQ-SF score <6
5. Patient has no erectile dysfunction (defined as IIEF-6 score ≥ 26)
6. Patient is willing to return for all visits as defined in the protocol
7. Patient is willing to follow the instruction of the Investigator
8. Patient has provided written informed consent

Exclusion Criteria:

1. Previous history of pelvic radiation
2. Previous history of simple prostatectomy or transurethral prostate surgery
3. Previous history of systemic therapy for prostate cancer
4. Patient has neurogenic bladder
5. Body weight less than 50 kg (110 pounds) or a body mass index greater than 40 kg/m2
6. History of open pelvic surgery within 5 years except for hernia repair
7. Scheduled at the time of screening to undergo chemotherapy, radiation, hormone therapy, or open surgery during the study period.
8. Any neurologic disorder or psychiatric disorder (e.g., Parkinson's Multiple Sclerosis, etc.) that might confound postsurgical assessments
9. Received administration of an investigational drug within 30 days prior to study, and/or has planned administration of another investigational product or procedure during participation in this study
10. Previous history of anaphylaxis or hypersensitivity to liposomal amphotericin- B

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients will be recruited as we are studying prostate cancer.
Enrollment: 100 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Erectile function | At three months post surgery
  Erectile function will be evaluated using the International Index of Erectile Function (IIEF)
Erectile function | At six months post surgery
  Erectile function will be evaluated using the International Index of Erectile Function (IIEF)
Erectile function | At twelve months post surgery
  Erectile function will be evaluated using the International Index of Erectile Function (IIEF)

SECONDARY OUTCOMES:
Potency endpoint | 6 weeks post op
  IIEF-6 Levels at 6 weeks post-op between the two treatment groups
Potency endpoint | 3 months post op
  IIEF-6 Levels at 3 months post-op between the two treatment groups
Potency endpoint | 6 months post op
  IIEF-6 Levels at 6 months post-op between the two treatment groups
Potency endpoint | 12 months post op
  IIEF-6 Levels at 12 months post-op between the two treatment groups
Return to continence | At 6 weeks post surgery
  Continence will be evaluated using the International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF)
Return to continence | At three months post surgery
  Continence will be evaluated using the International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF)
Return to continence | At six months post surgery
  Continence will be evaluated using the International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF)
Return to continence | At twelve months post surgery
  Continence will be evaluated using the International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF)
Pad Weight | 6 weeks post op
  Changes from baseline of average pad weight to 6 weeks post-op between treatment groups
Pad Count | 6 weeks post op
  Proportion of patients that wear 0 or 1 safety pads; 1-2 safety pads; and >2 safety pads per day
Pad Weight | 3 months post op
  Changes from baseline of average pad weight to 3 months post-op between treatment groups
Pad Count | 3 months post op
  Proportion of patients that wear 0 or 1 safety pads; 1-2 safety pads; and >2 safety pads per day
Pad Weight | 6 months post op
  Changes from baseline of average pad weight to 6 months post-op between treatment groups
Pad Count | 6 months post op
  Proportion of patients that wear 0 or 1 safety pads; 1-2 safety pads; and >2 safety pads per day
Pad Weight | 12 months post op
  Changes from baseline of average pad weight to 12 months post-op between treatment groups
Pad Count | 12 months post op
  Proportion of patients that wear 0 or 1 safety pads; 1-2 safety pads; and >2 safety pads per day
Sexual encounter | At three months post surgery
  Patients will be asked to complete the Sexual Encounter Profile (SEP) Diary to document after each sexual attempt
Sexual encounter | At six months post surgery
  Patients will be asked to complete the Sexual Encounter Profile (SEP) Diary to document after each sexual attempt
Sexual encounter | At twelve months post surgery
  Patients will be asked to complete the Sexual Encounter Profile (SEP) Diary to document after each sexual attempt
Biochemical recurrence endpoint | 6 weeks post-op
  Proportion of patients with biochemical recurrence at 6 weeks post-op between groups.
Biochemical recurrence endpoint | 3 months post-op
  Proportion of patients with biochemical recurrence at 3 months post-op between groups.
Biochemical recurrence endpoint | 6 months post-op
  Proportion of patients with biochemical recurrence at 6 months post-op between groups.
Biochemical recurrence endpoint | 12 months post-op
  Proportion of patients with biochemical recurrence at 12 months post-op between groups.
Patient intercourse satisfaction endpoint | 6 weeks post op
  Patient satisfaction using Likert score at 6 weeks post-op between groups
Patient intercourse satisfaction endpoint | 3 months post op
  Patient satisfaction using Likert score at 3 months post-op between groups
Patient intercourse satisfaction endpoint | 6 months post op
  Patient satisfaction using Likert score at 6 months post-op between groups
Patient intercourse satisfaction endpoint | 12 months post op
  Patient satisfaction using Likert score at 12 months post-op between groups
Failure Events of Following RARP endpoint | 2 weeks post-op
  Incidence of readmission for hospital stay at 2 weeks post-op between groups.
Failure Events of Following RARP endpoint | 2 weeks post-op
  Number of surgical interventions at 2 weeks post-op between groups

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stifelman, MD, Principal Investigator — Chair of Urology Department
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No